CLINICAL TRIAL: NCT00353171
Title: Organochlorine Exposure in Relation to Timing of Natural Menopause
Status: Completed | Type: Observational
Sponsor: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999903045; 03-E-N045
Record Dates: First submitted 2006-07-17; First posted 2006-07-18 (Estimated); Last update posted 2019-06-17 (Actual); Status verified 2019-05-29

CONDITIONS: Menopause
Keywords: Smoking; PCB; DDE; Menstrual Cycle; NC Infant Feeding Study
MeSH Terms: conditions — Smoking

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
This study will examine whether exposure to organochlorines (certain chemicals such as PCBs and DDE, used in pesticides or other industrial applications) is related to age at natural menopause. It is known, for example, that smokers experience menopause 1 to 2 years earlier than do non-smokers. This study will look for a similar association between organochlorine exposure and menopause. It will also look for possible associations between specific factors, such as pregnancy history and weight change, and changes over time in blood organochlorine levels.

Women who participated in the North Carolina Infant Feeding Study between 1978 and 1982 are eligible for this study. Participants will be interviewed over the phone for information about their reproductive and menstrual history, as well as additional information that may be related to age and menopausal status. Specifically, the interview will cover the following areas: 1) pregnancy and breastfeeding history; 2) menstrual periods and menopause; 3) use of birth control pills and hormone replacement therapy; 4) surgeries on the uterus or ovaries, such as hysterectomy or oophorectomy, or both; 5) smoking and alcoholic beverage consumption; 6) physical activity; 7) weight history; and 8) medical history. About one-half of the participants will have a blood sample drawn for analysis of the reproductive hormones FSH (follicle-stimulating hormone) and LH (leuteinizing hormone) and of DDE and PCB levels.

DETAILED DESCRIPTION:
Smoking has been shown in many studies to be associated with a 1-2 year decrease in age at natural menopause. However, relatively little is known about the effect of other potential toxicants, including organochlorines such as polychlorinated biphenyls (PCBs), and 1, 1 dichloro-2,2-bis(p-chlorophenyl) ethylene (p,p -DDE, referred to subsequently as DDE). We will assess timing of menopause among women who participated in the North Carolina Infant Feeding Study (total n = 865). Recruitment for this study was conducted between 1978 and 1982. PCB and DDE levels were analyzed in blood and breast milk samples around delivery and after pregnancy. The median age of the women as of March, 2002, is 50 years. Data will be collected in a telephone interview focusing on reproductive and menstrual history with additional information collected on demographic, social and behavioral factors that could affect timing of menopause. A blood sample will be collected from approximately 50% of participants based on sampling strata that involve criteria relating to age and menopausal status. Follicle stimulating hormone and luteinizing hormone will be measured in these samples in order to classify menopausal status of women who had undergone hysterectomy with retention of at least one ovary, women who are currently using hormone replacement therapy whose use began while still having periods, and women who report very short, very long, or irregular menstrual cycle lengths during the past 12 months. PCB and DDE levels will also be determined in these samples, allowing us to assess the correlation between current and baseline (1978-1982) PCB and DDE measures. The purpose of this study is to assess the association between the baseline organochlorine measurements and timing of natural menopause. A secondary aim will be to conduct exploratory analyses of the association between specific factors (e.g., pregnancy history, weight change) and rate of change in organochlorine levels.

ELIGIBILITY:
* INCLUSION AND EXCLUSION CRITERIA:

There will be no exclusions based on age, ethnicity or race/ethnicity. Participants who are unable to complete a telephone interview because of chronic illness (including cognitive impairment) or language or hearing difficulties will not be eligible.

There are 8 women in the cohort whose study children are known to have died. We will exclude these women from this follow-up study.

This leaves 857 women that are eligible for tracing the follow-up interview.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 514 (Actual)
Dates: Start 2003-03-01; Study Completion 2019-05-29

PRIMARY OUTCOMES:
Organochlorine & Nat. Menopause

SECONDARY OUTCOMES:
Rate of change of organochlorine levels

CONTACTS AND LOCATIONS:
Overall Officials: Donna D Baird, Ph.D., Principal Investigator — National Institute of Environmental Health Sciences (NIEHS)
Locations (1):
- NIEHS, Research Triangle Park, Research Triangle Park, North Carolina, United States

REFERENCES:
- [Background] McKinlay SM, Bifano NL, McKinlay JB. Smoking and age at menopause in women. Ann Intern Med. 1985 Sep;103(3):350-6. doi: 10.7326/0003-4819-103-3-350. PMID 4026083
- [Background] Cramer DW, Xu H. Predicting age at menopause. Maturitas. 1996 Apr;23(3):319-26. doi: 10.1016/0378-5122(96)00992-9. PMID 8794427
- [Background] Luoto R, Kaprio J, Uutela A. Age at natural menopause and sociodemographic status in Finland. Am J Epidemiol. 1994 Jan 1;139(1):64-76. doi: 10.1093/oxfordjournals.aje.a116936. PMID 8296776